CLINICAL TRIAL: NCT00825773
Title: A Randomized Study to Evaluate Safety and Efficacy of the ExcelTM Sirolimus Eluting Stent With a Biodegradable Polymer Versus SirOlimus ELUting Stent With Non-Biodegradable Polymer in the Treatment of PatIents With de nOvo Coronary Artery LesioNs
Brief Title: A Study to Evaluate Safety and Efficacy of the ExcelTM Sirolimus Eluting Stent With a Biodegradable Polymer Versus Sirolimus Eluting Stent With Non-Biodegradable Polymer in the Treatment of Patients With de Novo Coronary Artery Lesions
Acronym: EVOLUTION
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: JW Medical Systems Ltd (Industry)
Responsible Party: Yongzhi Yan, JW Medical Systems Ltd
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-09-01-19; ZSH-20090119
Record Dates: First submitted 2009-01-19; First posted 2009-01-21 (Estimated); Last update posted 2009-01-26 (Estimated); Status verified 2009-01

CONDITIONS: Ischemia; Cardiac Death; Myocardial Infarction
Keywords: TVF; TLF; MACE; Ischemia-driven Target Vessel Failure (TVF) at 12 months.; Ischemia-driven Target Lesion Failure (TLF) at 12 months defined as a; composite of cardiac death that can not be clearly attributed to a vessel; other than the target vessel, target vessel MI (Q and Non-Q wave) and; ischemia-driven TLR.; Rates of stent thrombosis, defined (per ARC definition) as definite or probable; and categorized as early, late or very late.; Major Adverse Cardiac Events (MACE) defined as cardiac death, target; vessel MI (Q and Non-Q wave), or target lesion revascularization (TLR) at 30; days, 6 months, 12 months and 2 to 5 years annually.
MeSH Terms: conditions — Ischemia; Death; Myocardial Infarction; Cardiovascular Diseases; Erythema Multiforme | interventions — Angioplasty, Balloon, Coronary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Excel (Active Comparator): Patients will be randomly assigned (2:1) to one of two treatment arms (the Excel DES or the Cypher DES). Randomization will be stratified by study site and number of vessels intended to be treated by the site investigator. Randomization will be accomplished through use of envelope randomization at the sites using the pre-assigned envelope randomization system. The study patient is considered enrolled upon randomization.
  Interventions: Device: Percutaneous Transluminal Coronary Angioplasty
- Cypher (Sham Comparator): Patients will be randomly assigned (2:1) to one of two treatment arms (the Excel DES or the Cypher DES). Randomization will be stratified by study site and number of vessels intended to be treated by the site investigator. Randomization will be accomplished through use of envelope randomization at the sites using the pre-assigned envelope randomization system. The study patient is considered enrolled upon randomization.
  Interventions: Device: Percutaneous Transluminal Coronary Angioplasty

INTERVENTIONS:
Device: Percutaneous Transluminal Coronary Angioplasty — Patients will be randomly assigned (2:1) to one of two treatment arms (the Excel DES or the Cypher DES). Randomization will be stratified by study site and number of vessels intended to be treated by the site investigator. Randomization will be accomplished through use of envelope randomization at the sites using the pre-assigned envelope randomization system. The study patient is considered enrolled upon randomization.
  Other Names: EVOLUTION; EXCEL vs CYPHER

SUMMARY:
E.V.O.L.U.T.I.O.N.: A Randomized Study to Evaluate Safety and Efficacy of the Excel Sirolimus Eluting Stent with a Biodegradable Polymer Versus Sirolimus Eluting Stent with a Non-Biodegradable Polymer in the Treatment of Patients with de novo Coronary Artery Lesions.

DETAILED DESCRIPTION:
E.V.O.L.U.T.I.O.N.: A Randomized Study to Evaluate Safety and Efficacy of the Excel Sirolimus Eluting Stent with a Biodegradable Polymer Versus Sirolimus Eluting Stent with a Non-Biodegradable Polymer in the Treatment of Patients with de novo Coronary Artery Lesions.

A prospective, randomized, controlled, parallel two-arm multi-center study, comparing the ExcelTM DES to CypherTM DES in the treatment of patients with de novo coronary artery lesions.

To evaluate the safety and efficacy of the Excel DES (biodegradable polymer) compared to the Cypher DES (non-biodegradable polymer) in the treatment of patients with de novo coronary artery lesions.

Approximately 1944 patients will be enrolled in up to 25 centers in China. Primary Endpoint:Ischemia-driven Target Vessel Failure which is a composite of cardiac death, myocardial infarction (Q and non-Q wave) and target vessel revascularization (TVR) at 12 months.

Secondary Endpoint:

1. Ischemia-driven Target Lesion Failure (TLF) at 12 months defined as a composite of cardiac death that can not be clearly attributed to a vessel other than the target vessel, target vessel MI (Q and Non-Q wave) and ischemia-driven TLR.
2. Rates of stent thrombosis, defined (per ARC definition) as definite or probable and categorized as early, late or very late.
3. Rates for each component of the TLF composite endpoint (cardiac death, target vessel MI, ischemia- driven TLR) at 12 months post-procedure.
4. Major Adverse Cardiac Events (MACE) defined as cardiac Death, target vessel MI (Q and Non-Q wave), or target Lesion revascularization (TLR) at 30 days, 6 months, 12 months and 2 to 5 years annually.
5. Device Success defined as achievement of a final residual in-stent diameter stenosis of < 30% (visual estimate) and a TIMI flow of 3 using the Excel/Cypher DES.
6. Procedure Success defined as achievement of a final in- stent diameter stenosis of < 30% (visual estimate) and a TIMI flow of 3 using any percutaneous method, without the occurrence of in-hospital MACE. (ALL TLR IN THIS STUDY WILL BE CLINICALLY INDICATED)

ELIGIBILITY:
Inclusion Criteria:

1. Patient > 18 years of age.
2. Diagnosis of stable angina, unstable angina or silent ischemia (evidence of myocardial ischemia).
3. Positive functional study or reversible change in the electrocardiogram (ECG) consistent with ischemia.
4. Patient must be an acceptable candidate for coronary artery bypass graft (CABG) surgery.
5. Patient must agree to undergo all required follow-up exam- inations.

Angiographic Inclusion Criteria:

1. Presence of one or more de novo coronary artery stenosis > 50% in native coronary arteries that corresponds with the evidence of ischemia. NOTE: In the presence of multiple de novo coronary lesions a maximum of four (4) planned Excel or Cypher stents may be used.
2. The target lesion(s) must be < 24mm in length and the reference diameter is > 2.5 mm and < 3.75 mm (visual estimate).

Exclusion Criteria:

1. Patient is pregnant or breast feeding.
2. Patient is allergic or has a contraindication to aspirin, clopidogrel and ticlopidine, heparin and bivalirudin, stainless steel, PLA, contrast media (that can not be adequately pre- medicated), and sirolimus (or its analogues).
3. Patient has evidence of an Acute Myocardial Infarction evidenced by elevation of CK/CK-MB or Troponin per clinical site standards, within 72 hours of the index procedure.
4. Patient is unable to provide informed consent.
5. Patient is participating in another device or drug study that has not reached the primary endpoint of the study.
6. Patient is considered for a DES other than the Excel or the Cypher stents.
7. Patient has a co-morbid condition(s) that could limit the patient's ability to participate in the study, comply with follow- up requirements and impact the scientific integrity of the study.

Angiographic Exclusion Criteria:

1. Patient has undergone previous stenting anywhere within the target vessel(s) within the previous 12 months, or will require stenting within the target vessel(s) within 12 months after the study procedure, or has received coronary brachytherapy at anytime.
2. Heavily calcified target lesion(s) which cannot be successfully pre-dilated.
3. Target lesion(s) involves a side branch >2.5 mm in diameter, or < 2.5 mm in diameter requiring treatment.
4. Patient has an unprotected Left Main Coronary Lesion with a diameter of >= 50%.
5. Anticipated use of rotoblator or cutting balloon on target lesion(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1944 (Estimated)
Dates: Start 2008-10; Primary Completion 2010-04 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Ischemia-driven Target Vessel Failure which is a composite of cardiac death, myocardial infarction (Q and non-Q wave) and target vessel revascularization (TVR) at 12 months. | 12 months

SECONDARY OUTCOMES:
Rates of stent thrombosis | 5 years
Rates for each component of the TLF composite endpoint at 12 months post-procedure | 5 years
Major Adverse Cardiac Events (MACE) at 30 days, 6 months, 12 months and 2 to 5 years annually | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- JW Medical Systems, Beijing, China

REFERENCES:
- [Background] Salam AM, Al Suwaidi J, Holmes DR Jr. Drug-eluting coronary stents. Curr Probl Cardiol. 2006 Jan;31(1):8-119. doi: 10.1016/j.cpcardiol.2005.09.002. PMID 16389102